CLINICAL TRIAL: NCT00046241
Title: A 7 Month, Multicenter, Randomized, Double-blind, Placebo-controlled Comparison of 150-300mg/Day of Extended-release Bupropion Hydrochloride and Placebo for the Prevention of Seasonal Affective Disorder in Subjects With a History of Seasonal Affective Disorder Followed by an 8-week Observational Follow-up Phase
Brief Title: Prevention of Seasonal Affective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK130930
Record Dates: First submitted 2002-09-24; First posted 2002-09-25 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Seasonal Affective Disorder
Keywords: seasonal depression winter blues winter depression
MeSH Terms: conditions — Seasonal Affective Disorder

INTERVENTIONS:
Drug: Extended-release bupropion hydrochloride

SUMMARY:
This is a placebo controlled study evaluating the effectiveness of medication in preventing depressive episodes in subjects with a history of Seasonal Affective Disorder (SAD).

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of Major Depressive Disorder (MDD) with a seasonal pattern.

Exclusion Criteria:

* Patient has a current or past history of seizure disorder or brain injury.
* Patient has a history or current diagnosis of anorexia nervosa or bulimia.
* Patient has recurrent summer depression more frequently than winter depression.
* Patient has primary diagnosis of panic disorder, Obsessive Compulsive Disorder (OCD), Posttraumatic Stress Disorder (PTSD), acute distress disorder, bipolar II disorder or other psychotic disorders.
* Patient has initiated psychotherapy within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-09 (Actual); Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Time between randomization and onset of a seasonal depressive episode. Proportion of depression-free subjects.

SECONDARY OUTCOMES:
Change in HAMD-24 and -17 total score. Change in pain score.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trial, MD, Study Director — GlaxoSmithKline
Locations (47):
- United States (40):
  - GSK Clinical Trials Call Center, Anchorage, Alaska
  - GSK Clinical Trials Call Center, Hamden, Connecticut
  - GSK Clinical Trials Call Center, Boise, Idaho
  - GSK Clinical Trials Call Center, Chicago, Illinois
  - GSK Clinical Trials Call Center, Edwardsville, Illinois
  - GSK Clinical Trials Call Center, Oak Brook, Illinois
  - GSK Clinical Trials Call Center, Oakbrook Terrace, Illinois
  - GSK Clinical Trials Call Center, Lafayette, Indiana
  - GSK Clinical Trials Call Center, Cedar Rapids, Iowa
  - GSK Clinical Trials Call Center, Overland Park, Kansas
  - GSK Clinical Trials Call Center, Baltimore, Maryland
  - GSK Clinical Trials Call Center, Rockville, Maryland
  - GSK Clinical Trials Call Center, Belmont, Massachusetts
  - GSK Clinical Trials Call Center, Detroit, Michigan
  - GSK Clinical Trials Call Center, Farmington Hills, Michigan
  - GSK Clinical Trials Call Center, Minneapolis, Minnesota
  - GSK Clinical Trials Call Center, St Louis, Missouri
  - GSK Clinical Trials Call Center, Omaha, Nebraska
  - GSK Clinical Trials Call Center, Clementon, New Jersey
  - GSK Clinical Trials Call Center, Kenilworth, New Jersey
  - GSK Clinical Trials Call Center, Princeton, New Jersey
  - GSK Clinical Trials Call Center, Albany, New York
  - GSK Clinical Trials Call Center, New York, New York
  - GSK Clinical Trials Call Center, Rochester, New York
  - GSK Clinical Trials Call Center, Beachwood, Ohio
  - GSK Clinical Trials Call Center, Cincinnati, Ohio
  - GSK Clinical Trials Call Center, Dayton, Ohio
  - GSK Clinical Trials Call Center, Marion, Ohio
  - GSK Clinical Trials Call Center, Eugene, Oregon
  - GSK Clinical Trials Call Center, Portland, Oregon
  - GSK Clinical Trials Call Center, Havertown, Pennsylvania
  - GSK Clinical Trials Call Center, Jenkintown, Pennsylvania
  - GSK Clinical Trials Call Center, Philadelphia, Pennsylvania
  - GSK Clinical Trials Call Center, East Providence, Rhode Island
  - GSK Clinical Trials Call Center, Woodstock, Vermont
  - GSK Clinical Trials Call Center, Falls Church, Virginia
  - GSK Clinical Trials Call Center, Bellevue, Washington
  - GSK Clinical Trials Call Center, Seattle, Washington
  - GSK Clinical Trials Call Center, Spokane, Washington
  - GSK Clinical Trials Call Center, Brown Deer, Wisconsin
- Canada (7):
  - GSK Clinical Trials Call Center, Calgary, Alberta
  - GSK Clinical Trials Call Center, Edmonton, Alberta
  - GSK Clinical Trials Call Center, Kelowna, British Columbia
  - GSK Clinical Trials Call Center, Winnipeg, Manitoba
  - GSK Clinical Trials Call Center, Toronto, Ontario
  - GSK Clinical Trials Call Center, Montreal, Quebec
  - GSK Clinical Trials Call Center, Sherbrooke, Quebec